CLINICAL TRIAL: NCT04050228
Title: A Phase II Study of Quantitative Ultrasound to Guide Adaptive Chemotherapy Among Women With Locally Advanced Breast Cancer (LABC)
Brief Title: Use of Quantitative Ultrasound to Guide Adaptive Chemotherapy Among Women With Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Gregory Czarnota, Radiation Oncologist and Clinician Scientist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 308-2017
Record Dates: First submitted 2019-07-22; First posted 2019-08-08 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer
Keywords: Ultrasound, Chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The trial design is a Phase II study to demonstrate the use of quantitative ultrasound to guide adaptive chemotherapy for patients with breast cancer. The primary endpoint will be measurement of improved response rate locally. Patients were randomly allocated in 1:1 ratio to a standard arm or experimental arm stratified by hormonal receptor status
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Neoadjuvant Chemotherapy Monitoring (No Intervention): Patients who will be randomized to the control arm with Standard Neoadjuvant Chemotherapy Monitoring will receive Phase I chemotherapy consisting of anthracycline-based treatment followed by Phase II chemotherapy consisting of taxane-based treatment.
  Patients will be imaged but no modifications to treatment will occur in this trial arm depending on response by quantitative ultrasound.
- Adaptive Chemotherapy Monitoring (Experimental): Patients who will be randomized to the experimental arm Adaptive Chemotherapy Monitoring and demonstrate Response (+) will continue until standard chemotherapy is completed. For patients who do not demonstrate response after 4 weeks of chemotherapy, an early switch to the second phase of chemotherapy could occur (Phase II/Taxane) At the discretion of the treating medical oncologist.
  Patients will undergo Quantitative Ultrasound on the following time points: Pre-treatment, Weeks 1, 4, 8, 12 and Pre-Operatively. These QUS time points correspond to the following chemotherapy times.
  Interventions: Device: Quantitative ultrasound to guide adaptive chemotherapy

INTERVENTIONS:
Device: Quantitative ultrasound to guide adaptive chemotherapy — Quantitative ultrasound results will be used to measure chemotherapy response and guide an adaptive chemotherapy strategy for patients who are found to be nonresponders to their chemotherapy.
  Arms: Adaptive Chemotherapy Monitoring

SUMMARY:
The primary objective of this study is to assess the feasibility of randomizing breast cancer patients to quantitative ultrasound to guide adaptive Neoadjuvant Chemotherapy as compared to standard clinical monitoring and therapy. The Investigators have previously demonstrated that high-frequency ultrasound and spectroscopy, and recently conventional-frequency ultrasound and spectroscopy may be used to detect cell death in vitro, in situ and in vivo. The method can detect different forms of cell death and has been demonstrated to be sensitive to apoptotic, necrotic and mitotic cell death. By detecting cell death early in a treatment on the order of hours to days, rather than traditional anatomical assessments that take place weeks to months after the completion of therapy, ineffective therapies could be switched to more efficacious treatments or aggressive salvage therapy which has shown to already benefit patients. The overarching goal of this research is to transform the delivery of neoadjuvant chemotherapy using quantitative ultrasound (QUS), which is non-invasive, inexpensive and portable.

DETAILED DESCRIPTION:
This study phase II will demonstrate the use of quantitative ultrasound to guide adaptive chemotherapy for patients with breast cancer. The primary endpoint will be measurement of improved response rate locally. This trial will enroll 240 randomized breast cancer patients to be assess with quantitative ultrasound to guide adaptive neoadjuvant chemotherapy as compared to standard clinical monitoring and therapy. We will evaluate the safety of its use and expect equivalence in this small patient population. This will allow for more accurate estimation of a needed sample size for a phase III superiority trial.

ELIGIBILITY:
Inclusion Criteria:

1. Women ≥ 18 years of age
2. Diagnosis of breast cancer with a primary tumour >2cm in size
3. With conditions meeting criteria for chemotherapy administration
4. Normal hematological blood counts (hemoglobin ≥ 100 g/l, platelet count ≥ 100 x 109, absolute neutrophil count ≥ 2.0 x109 cells per L)
5. Creatinine ≤175 µmol/L
6. Liver enzymes (AST and ALT) ≤ 1.5 times upper limit of normal
7. Cardiac function (left ventricular ejection fraction) ≥55%
8. Eligible for neoadjuvant chemotherapy.

Exclusion Criteria:

1. Inflammatory breast cancer
2. Contraindications to neoadjuvant treatment including pregnancy or lactation
3. Past medical history of connective tissue disease
4. Past history of dermatologic disease involving the breast
5. Eastern Cooperative Group Status (ECOG) ≥3
6. No peripheral neuropathy of a severity of grade ≥2
7. Evidence of distant metastatic disease
8. Known sensitivity to components present in ultrasound gel.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women ≥ 18 years of age with breast cancer eligible for neoadjuvant chemotherapy
Enrollment: 240 (Estimated)
Dates: Start 2018-06-13 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Measuring the rate of treatment response between the treatment groups | Up to 5 years
  To assess the feasibility of randomizing breast cancer patients to quantitative ultrasound to guide adaptive neoadjuvant chemotherapy as compared to standard clinical monitoring and therapy.

SECONDARY OUTCOMES:
Clinical efficacy of quantitative ultrasound | Up to 5 years
  Sensitivity and specificity of quantitative ultrasound will be calculated against surgical pathologic response documented after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory J Czarnota, PhD, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Moore-Palhares D, Alberico D, Chan AW, DiCenzo D, Sannachi L, Dasgupta A, Yip J, Pena MLA, Gandhi S, Pezo R, Eisen A, Jerzak KJ, Gonzalez CAC, Warner E, Wright FC, Look-Hong N, Roberts A, Sadeghi-Naini A, Curpen B, Skarpathiotakis M, Betel C, Kolios MC, Trudeau M, Czarnota GJ. Quantitative ultrasound imaging for predicting response and guiding personalized neoadjuvant chemotherapy in breast cancer: randomized phase 2 clinical trial results. NPJ Precis Oncol. 2025 Dec 4;9(1):390. doi: 10.1038/s41698-025-01134-x. PMID 41345775
- [Derived] Dasgupta A, DiCenzo D, Sannachi L, Gandhi S, Pezo RC, Eisen A, Warner E, Wright FC, Look-Hong N, Sadeghi-Naini A, Curpen B, Kolios MC, Trudeau M, Czarnota GJ. Quantitative ultrasound radiomics guided adaptive neoadjuvant chemotherapy in breast cancer: early results from a randomized feasibility study. Front Oncol. 2024 Apr 19;14:1273437. doi: 10.3389/fonc.2024.1273437. eCollection 2024. PMID 38706611